CLINICAL TRIAL: NCT02900677
Title: Developing and Testing the Effects of Patient-centered Prehabilitation Program on Improving Fatigue, Nutritional Status, and Quality of Life in Patients With Operable Pancreatic Cancer Perioperatively and Following Surgery
Brief Title: Developing Prehabilitation Program in Patients With Operable Pancreatic Cancer Perioperatively and Following Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201505160RINB
Record Dates: First submitted 2016-08-24; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Fatigue; Nutrition; Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms; Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical and nutrition program (Experimental): 6 education programs with physical enhancement and nutrition related information for 12 weeks.
  Interventions: Behavioral: Physical and nutrition program
- Control (No Intervention): usual care

INTERVENTIONS:
Behavioral: Physical and nutrition program — 6 education programs with physical enhancement and nutrition related information for 12 weeks
  Arms: Physical and nutrition program

SUMMARY:
The aims of this three-year study are to:

1. explore the change of fatigue, nutritional status, quality of life and care needs in patients with operable pancreatic cancer perioperatively and following surgery within 3 months.
2. develop and evaluate the effect of patient-centered cancer prehabilitation care program on improving fatigue, nutritional status and quality of life (QOL) in this population.

DETAILED DESCRIPTION:
Develop and evaluate the effect of patient-centered cancer prehabilitation care program on improving fatigue, nutritional status and quality of life (QOL) in this population.

ELIGIBILITY:
Inclusion Criteria:

* patients with pancreatic cancer and are going to receive surgery.

Exclusion Criteria:

* poor functional status

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Self-report Questionnaire | Change from baseline physical symptom at 12 months
  The questionnaire includes 25 items to assess the physical symptom distresses

SECONDARY OUTCOMES:
Self-report Questionnaire | Change from baseline fatigue at 12 months
  The questionnaire includes 14 items to assess fatigue intensity and duration

OTHER OUTCOMES:
Self-report Questionnaire | Change from baseline quality of life at 12 months
  The questionnaire includes 32 items to assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PHD, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang HY, Shun SC, Lee YH, Liou YT, Chou YJ, Kuo HJ, Tien YW, Lai SR, Hung H. Trajectories of perioperative nutritional status in patients with pancreatic tumor after surgery in six months. Eur J Oncol Nurs. 2024 Oct;72:102687. doi: 10.1016/j.ejon.2024.102687. Epub 2024 Aug 21. PMID 39288676